CLINICAL TRIAL: NCT00199264
Title: A Single-Blind, Randomized, Dose-Finding Study Versus Fluconazole to Assess the Efficacy and Tolerability of Five Single Doses of Albaconazole in the Treatment of Acute Non-Recurrent Candida Spp Vulvovaginitis
Brief Title: Efficacy Vulvovaginitis Candida
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: J. Uriach and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICO8ATM/2/03
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2003-10

CONDITIONS: Candidiasis Vulvaginitis
Keywords: antifungal oral therapy; efficacy acute candidiasis vulvaginitis
MeSH Terms: interventions — albaconazole

INTERVENTIONS:
Drug: Albaconazole oral solution

SUMMARY:
To compare the therapeutic efficacy of 10 mg, 40 mg, 80 mg, 160 mg and 320 mg of albaconazole, as a single oral dose, in women affected by acute non-complicated vulvovaginitis due to Candida spp.

DETAILED DESCRIPTION:
Multi-center, open-label, randomized study, controlled with fluconazole.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients over 18 years of age, with a vaginal score sum ³ 2 and KOH fresh examination positive for yeasts (hyphae, pseudohyphae). The diagnosis must be later confirmed with a positive Candida spp. culture.

Exclusion Criteria:

* Patients with recurrent disease, prior treatment with antifungal agents within the last 7 days, immunosuppression, pregnant or lactating women, other vulvovaginal diseases, other systemic diseases, hypersensitivity to azole derivatives.Number of patients: 78 patients included to obtain 60 evaluable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-06; Study Completion 2004-10

PRIMARY OUTCOMES:
Primary Efficacy VariableThe primary efficacy assessment will be carried out 24 ± 4 (FV) days following treatment or at the last patient's.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Negroni, Dr, Study Chair — Hosp Infecciosas F J Muñiz, Buenos Aires. Argentina